CLINICAL TRIAL: NCT05048888
Title: Symphony IL-6 Reference Range Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bluejay Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CES-0001
Record Dates: First submitted 2021-09-09; First posted 2021-09-17 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Symphony IL-6 is a device that quantitates human IL-6 by fluorescence enzyme immunoassay (FEIA) from whole-blood specimens. Use of Symphony IL- 6 removes the need for plasma separation before testing. Symphony IL-6 comprises two components, the Symphony Fluorescence Immunoanalyzer and the Symphony IL-6 Cartridge. Whole blood is added to the cartridge and then up to six cartridges can be inserted into the immunoanalyzer. After 20 minutes a readout and printout are given with a quantitative IL-6 concentration. The used cartridges are fully enclosed and can be easily disposed of in general hospital bio-waste. Given the nature of this device and its portability, there is potential for future deployment as a point-of-care (POC) device.

The objective of this study is to establish a reference range for Symphony IL-6 in a cohort of apparently healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to provide informed consent
* > 18 years of age
* Whole blood specimen collected in EDTA anticoagulant tubes
* Minimum volume of 100µL for Symphony IL-6 testing
* Specimen is available for testing within 12 hours from collection
* C-Reactive Protein (CRP) < 10 mg/L

Exclusion Criteria:

* Subjects presenting with a fever
* Subjects with a diagnosis of COVID-19 or other respiratory illness at the time of collection
* Subjects otherwise self-reported as unhealthy
* Hemolyzed specimens

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will enroll approximately 120 apparently healthy individuals, split approximately between males and females, and covering an age range from approximately 18 to 85 years of age at the University of Texas Southwestern Medical Center, or from satellite facilities associated with the medical center. Subjects must meet all eligibility criteria to be in enrolled in the study. Whole blood specimens will be prospectively collected and tested using the Symphony IL-6 system.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
IL-6 Reference Range Study | Specimen is tested within 12 hours from collection
  Establishment of the interleukin-6 concentration in whole blood samples from healthy individuals.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States